CLINICAL TRIAL: NCT05172401
Title: A Multi-Center, Open-label, 24-week Clinical Investigation to Evaluate Safety and Tolerability of Treatment With the Oxulumis®, Suprachoroidal Drug Administration Device Delivering 2.4mg Triesence® With Diabetic Macular Edema
Brief Title: Oxulumis®, Suprachoroidal Drug Administration of Triesence® in Diabetic Macular Edema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unforeseen, continued (>12month) global shortage of study medication. Study Drug Triesence, manufacturer Novartis, not supplied throughout 2022
Sponsor: Oxular Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXUCT-101
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes Mellitus; Diabetic Retinopathy; Microcatheter; Suprachoroidal drug delivery; Clinical Investigation; Triamcinolone; Triamcinolone acetonide; Choroid; Suprachoroidal microcatheterization; Recalcitrant Macular Edema; Illuminated Microcatheter; Precision Drug Delivery
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Single-arm, single-dose, open-label, multi-center clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active Treatment - Oxulumis® - Triesence® (Experimental): The Oxulumis® device will be used for the administration of Triesence® (Triamcinolone acetonide) via suprachoroidal microcatheterization
  Interventions:
  * Device: Oxulumis® suprachoroidal microcatheterization device
  * Drug: Triesence® (Triamcinolone acetonide)
  Interventions: Device: Oxulumis® suprachoroidal microcatheterization administration of Triesence®

INTERVENTIONS:
Device: Oxulumis® suprachoroidal microcatheterization administration of Triesence® — Suprachoroidally administered Triamcinolone acetonide (Triesence) 2.4mg/60µl

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and tolerability of using the Oxulumis® microcatheterization device to administer Triesence® to the suprachoroidal space in participants with DME.

DETAILED DESCRIPTION:
This 24-week, single-arm, single-dose clinical investigation will evaluate the safety and tolerability and explore the efficacy of the Oxulumis® microcatheterization device to administer Triesence® (triamcinolone acetonide suspension) 2.4 mg to the posterior suprachoroidal space in subjects with DME not responding to standard therapy.

After a screening period, approximately 20 eligible subjects will receive a single dose of 2.4 mg Triesence® to the posterior suprachoroidal space.

The follow-up period after treatment administration will be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 1 or Type 2 diabetes mellitus.
* Have Diabetic Macular Edema (DME) involving the center of the fovea in the study eye with a central retinal thickness (CRT), at the screening visit, of≥ 320 for males or ≥ 305 for females on Spectralis (Heidelberg) or ≥ 305 for males or ≥ 290 for females with Cirrus (Zeiss) by spectral domain optical coherence tomography (SD-OCT).
* Have a best-corrected visual acuity (BCVA) in the study eye between 34 and 68 letters ETDRS at the screening visit.
* Have shown limited response to previous IVT treatment with anti-vascular endothelial growth factor (VEGF) agents or local corticosteroid treatment (IVT, subtenon, topical) defined as less than 20% reduction of central subfield thickness (CST) with previous treatments.
* Study eye suitable for suprachoroidal injection in the investigator's judgment in agreement with the medical monitor. Patients with ocular hypotony or structural abnormalities like choroidal coloboma or chorioretinal anastomosis, amongst others, are not eligible.

Exclusion Criteria:

* Presence of any other ocular condition in the study eye such that visual acuity may not improve from the resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, or nonretinal causes).
* Active proliferative diabetic retinopathy (PDR) or sequelae of PDR (including iris neovascularization, vitreous hemorrhage, or tractional retinal detachment) at screening in the study eye.
* Pan-retinal photocoagulation (PRP) or macular laser photocoagulation in the study eye performed within sixteen (16) weeks before screening.
* Prior IVT treatment with anti-VEGF in the study eye: last injection with ranibizumab or bevacizumab within four (4) weeks, aflibercept or brolucizumab within eight (8) weeks, faricimab within twelve (12) weeks before screening
* Prior ocular treatment with steroids in the study eye: last injection (intra- or periocular) with triamcinolone acetonide within three (3) months, with dexamethasone implant (Ozurdex®) within six (6) months before screening.
* Prior treatment with longer duration steroid implants (e.g., fluocinolone acetonide IVT implant, Iluvien®) is not allowed.
* Prior treatment with suprachoroidal steroids is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of ocular adverse events, systemic adverse events, serious, and treatment-emergent non-serious adverse events | 24 Weeks
  Treatment-emergent adverse events are defined as an event that emerges following administration of Triesence with the Oxulumis microcatheter administered at Visit 2 (Baseline, Day 0)
Frequency of adverse device effects and frequency of serious adverse device effects | 24 Weeks
  Adverse device effects and serious adverse device effects are defined as effects that emerge following the administration of the Oxulumis microcatheter at Visit 2 (Baseline, Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Asmus, MD, Study Director — Oxular Limited

IPD SHARING:
Plan to Share IPD: No